CLINICAL TRIAL: NCT03255434
Title: LEAn Body Mass Normalization of OXaliplatin Based Chemotherapy for Stage III Colon Cancer Patients Treated in Adjuvant Setting: Impact on Oxaliplatin-induced Sensitive Neurotoxicity. A Multicenter Phase II Randomized Trial (LEANOX)
Brief Title: LEAn Body Mass Normalization of OXaliplatin Based Chemotherapy
Acronym: LEANOX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICM-URC2016/27
Record Dates: First submitted 2017-08-11; First posted 2017-08-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stage III Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folfox 4 (Active Comparator): Standard FOLFOX4: Oxaliplatin and simplified LV5FU2 Dose of oxaliplatin 85mg/m²
  Interventions: Drug: Oxaliplatin
- Folfox 4 LBM (Experimental): Adapted FOLFOX4: Oxaliplatin and simplified LV5FU2 Dose of oxaliplatin allocated according to lean body mass (LBM)
  Interventions: Drug: Oxaliplatin LBM

INTERVENTIONS:
Drug: Oxaliplatin — Simplified FOLFOX 4 regimen: Association of Oxaliplatin (85 mg/m² ) + simplified LV5FU2 Length of a cycle : 2 days Interval between 2 cycles : 2 weeks (D1=D15) Expected number of cycles: 12
  Arms: Folfox 4
Drug: Oxaliplatin LBM — Simplified FOLFOX 4 regimen: Association of Oxaliplatin (LBM) + simplified LV5FU2
  Other Names: Oxaliplatin
  Arms: Folfox 4 LBM

SUMMARY:
Cytotoxic chemotherapy is usually scaled to the body surface area (BSA), and is currently not adjusted to the body proportions of lean and fat (i.e. body composition) of individual patients. Patients with low muscle mass behave like patients "overdosed" with chemotherapy resulted in dose-limiting toxicities (e.g. dose reductions, treatment delays or permanent treatment discontinuation), independently of the patient's weight.

DETAILED DESCRIPTION:
Adjuvant chemotherapy with fluoropyrimidines and Oxaliplatin is the current worldwide standard of care for stage III colorectal cancer (CRC). This regimen leads to significant cost, toxicity, and patient inconvenience. Oxaliplatin induces two distinct forms of neuropathy: a common acute syndrome that is transient (dysesthesia, contractures and numbness) and a dose-limiting chronic sensory neurotoxicity that is cumulative. Neurotoxicity is common; it affects 80% of patients and becomes chronic in 15-20% of cases, sometimes irreversibly. Chronic neurotoxicity can severely affect everyday life activities. To date, neuromodulators agents have failed to prevent neurotoxicity and Stop & Go strategies, intended to decrease the cumulative dose of Oxaliplatin administrated, are more appropriate for palliative treatment of advanced CRC. Recent data support the plausibility of a shorter duration of adjuvant treatment without loss of efficacy. This hypothesis is tested in several international trials.

Cytotoxic chemotherapy is usually scaled to the body surface area (BSA), and is currently not adjusted to the body proportions of lean and fat (i.e. body composition) of individual patients. The impact of body composition on drug metabolism is however well known: i.e. anesthetics accumulate in adipose tissue and specific precautions are essential to avoid overdose. Concerning chemotherapies, the lean body mass (LBM) may be the salient feature defining drug metabolism. A theme is emerging from recent studies: in patients with breast cancer and treated with 5-FU (whose dosage was calculated from the body surface), severe depletion of the LBM is a powerful predictor of excessive toxicity. Indeed, depletion of the LBM, as precisely defined by computed tomography, is a unique predictor of clinically unacceptable toxicity. Low LBM was shown to be a significant predictor of dose-limiting toxicity (DLT) in CRC patients administered 5-FU using a conventional BSA-based dosing and DLT was concentrated in patients receiving >20 mg 5FU/kg LBM. Two cohorts of CRC patients treated with Oxaliplatin showed that overall DLTs, and specifically Oxaliplatin-due neuropathy, occurred mostly in patients who receive > 3.09 mg/Oxaliplatin/kg LBM. Although, preliminary findings are available in hepatocellular carcinoma, the area under the concentration time curve (AUC) of Sorafenib cancer therapy was doubled in patients with depleted LBM (102.4 vs. 53.7ng/mL.h), which seem of interest. Patients with low muscle mass behave like patients "overdosed" with chemotherapy resulted in dose-limiting toxicities (e.g. dose reductions, treatment delays or permanent treatment discontinuation), independently of the patient's weight.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 18 years old up to 75 years old including. Histologically confirmed adenocarcinoma of the colon.
* Has undergone a curative resection for stage III colon cancer.
* Scheduled to receive 6 months of Oxaliplatin-based adjuvant chemotherapy at a dose of 85 mg/m² of Oxaliplatin every 2 weeks (simplified FOLFOX 4 regimen).
* The following laboratory values obtained ≤ 28 days prior to inclusion:

WBC ≥ 3000/mm3; ANC ≥1500/mm3; PLT ≥100,000/mm3; HgB ≥10.0g/dl; Total bilirubin ≤1.5 x upper normal limit (UNL); Serum creatinine ≤1.5 x UNL; Serum calcium ≤ 1.2 x UNL; Serum magnesium ≤ 1.2 x UNL.

* Central venous access line present or patient scheduled to have a central line placed prior to starting chemotherapy or the treatment protocol.
* Negative pregnancy test (serum or urine) done ≤ 7 days prior to registration, for women of childbearing potential only.
* Ability to complete questionnaire(s) by themselves or with assistance.
* ECOG Performance Status (PS) of 0, 1 for patients until 70 years old included and ECOG PS of 0 for patients between 70 to 75 years old included.
* Has provided informed written consent.
* Patient willing to provide blood sample for research purposes
* Patient affiliated to a French social security system

Exclusion Criteria:

* Pregnant or breastfeeding women
* Men or women of childbearing potential who are unwilling to employ adequate contraception since this study involves agents that have known genotoxic, mutagenic and teratogenic effects
* Pre-existing peripheral neuropathy of any grade.
* Prior treatment with neurotoxic chemotherapy such as Oxaliplatin, cisplatin, taxanes, or vinca alkaloids.
* Treatment with 1) the anticonvulsants carbamazepine (e.g., Tegretol®), phenytoin (e.g., Dilantin®), valproic acid (e.g. Depakine®), gabapentin (Neurontin®); pregabalin (Lyrica®); 2) the following neurotropic agents: venlafaxine (Effexor®), desvenlafaxine (Pristiq®), milnacipran (Savella®) or duloxetine (Cymbalta®); 3) Tricyclic antidepressants (such as amitryptilline) or 4) any other agent specifically given to prevent or treat neuropathy.
* Family history of a genetic/familial neuropathy.
* Participation in another medication trial within 30 days prior to study entry
* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to sign the informed consent or to terminate the study
* History of other solid tumor in 3 years before the inclusion, excepted of cancer in situ of the cervix and skin cancer (basal or squamous cell) treated and controlled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of neurotoxicity associated with Oxaliplatin | through study completion, an average of 5 years
  Neurotoxicity assessment

CONTACTS AND LOCATIONS:
Overall Officials: marc YCHOU, Study Director — Institut régional du Cancer de Montpellier
Locations (11):
- France (11):
  - Hôpital Européen, Marseille, Bouches Du Rhône
  - Centre hospitalier régional et universitaire de Montpellier, Montpellier, Hérault
  - CHU de Nancy, Vandœuvre-lès-Nancy, Lorraine
  - Insitut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe-et-Moselle,
  - Hôpital Saint-Jean, Perpignan, Pyrénées-orientales
  - Centre François Baclesse, Caen
  - CHU La TIMONE, Marseille
  - Institut regional du Cancer - Val d Aurelle, Montpellier
  - AP-HP Hôpital Saint-Louis, Paris
  - Centre Eugène Marquis, Rennes
  - Centre Paul Strauss, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Assenat E, Ben Abdelghani M, Gourgou S, Perrier H, Akouz FK, Desgrippes R, Galais MP, Janiszewski C, Mazard T, Rinaldi Y, Lepage C, Tetreau R, Senesse P. Impact of Lean Body Mass-Based Oxaliplatin Dose Calculation on Neurotoxicity in Adjuvant Treatment of Stage III Colon Cancer: Results of the Phase II Randomized LEANOX Trial. J Clin Oncol. 2025 Aug 10;43(23):2616-2627. doi: 10.1200/JCO-24-02754. Epub 2025 Jun 20. PMID 40540704